CLINICAL TRIAL: NCT00195897
Title: Early Assessment of Anthracycline-induced Cardiotoxicity: Usefulness of Biochemical Markers and Ventricular Function Assessment.
Brief Title: Early Assessment of Anthracycline-induced Cardiotoxicity (CARDIOTOX)
Status: Terminated | Type: Observational
Why Stopped: No patients; only 6 enrolled after 2 years
Sponsor: Centre Henri Becquerel (Other)
Collaborators: Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-001-CHB
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Lymphoma; Heart Failure, Congestive
Keywords: Lymphoma; Anthracyclines; Heart Failure; Radionuclide; Magnetic Resonance Imaging; Troponin; Natriuretic Peptide, Brain
MeSH Terms: conditions — Lymphoma; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Anthracycline-based chemotherapy is a key point of the treatment of patients with Hodgkin's and non-Hodgkin's lymphomas. However, cumulative doses are limited by cardiotoxicity, resulting in a marked left ventricular function impairment that may lead to heart failure.

The standard clinical approach to monitoring for anthracycline cardiotoxicity is based on cardiac function monitoring using echocardiography or radionuclide angiography. The aim of this study is to evaluate the usefulness of biochemical markers of cardiac injury (troponin and NT-proBNP) and structural changes on cardiac MR in predicting anthracycline cardiotoxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven lymphoma (Hodgkin's or non-Hodgkin's)
* Age > 18 y/o and < 70 y/o
* WHO score < or = 2
* Life expectancy > 6 mo
* Left ventricular ejection fraction > 50%
* Informed consent

Exclusion Criteria:

* Previous chemotherapy using anthracyclines
* History of radiation therapy
* History of congestive heart failure
* History of chronic renal insufficiency
* Contra indication to MR examination
* Atrial fibrillation and significant arrhythmia
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hodgkin lymphoma disease
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2006-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alain Manrique, MD, Study Chair — Centre Henri Becquerel; Fabrice Jardin, MD, Principal Investigator — Centre Henri Becquerel
Locations (2):
- France (2):
  - University Hospital of Rouen, Rouen
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardinale D, Sandri MT, Martinoni A, Borghini E, Civelli M, Lamantia G, Cinieri S, Martinelli G, Fiorentini C, Cipolla CM. Myocardial injury revealed by plasma troponin I in breast cancer treated with high-dose chemotherapy. Ann Oncol. 2002 May;13(5):710-5. doi: 10.1093/annonc/mdf170. PMID 12075738
- [Background] Singal PK, Iliskovic N. Doxorubicin-induced cardiomyopathy. N Engl J Med. 1998 Sep 24;339(13):900-5. doi: 10.1056/NEJM199809243391307. No abstract available. PMID 9744975
- [Background] Okumura H, Iuchi K, Yoshida T, Nakamura S, Takeshima M, Takamatsu H, Ikeno A, Usuda K, Ishikawa T, Ohtake S, Matsuda T. Brain natriuretic peptide is a predictor of anthracycline-induced cardiotoxicity. Acta Haematol. 2000;104(4):158-63. doi: 10.1159/000046508. PMID 11279304
- [Background] Mitani I, Jain D, Joska TM, Burtness B, Zaret BL. Doxorubicin cardiotoxicity: prevention of congestive heart failure with serial cardiac function monitoring with equilibrium radionuclide angiocardiography in the current era. J Nucl Cardiol. 2003 Mar-Apr;10(2):132-9. doi: 10.1067/mnc.2003.7. PMID 12673177